CLINICAL TRIAL: NCT05677698
Title: Menoupausal Symptoms and Aromatherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Karatayhfz
Record Dates: First submitted 2022-11-16; First posted 2023-01-10 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-11

CONDITIONS: Aromatherapy
Keywords: aromatherapy; menopause
MeSH Terms: interventions — lemon oil; peppermint oil; almond oil

STUDY DESIGN:
Intervention Model Description: Massage will be done for 4 weeks and 2 times a week (8 massages will be given to a person in total). Experimental groups: The researcher will add 2 drops of aromatic oil to 5 cc almond oil and give hand and arm massage to the participants for 30 minutes. Peppermint oil will be used in the first experimental group, lemon oil in the second experimental group and only almond oil in the control group. The fragrance to be used before starting the application will be given to the women by giving them a sniff.Placebo Group: Hand and arm massage will be performed for 30 minutes by the researcher using only almond oil. Three groups will be formed from women with menopausal symptoms. 1st group will be given a massage with Mint, 2nd group Lemon, 3rd group (placebo group-almond oil) and menopausal symptoms, happiness, peace and aging anxiety symptoms will be evaluated between the groups. All groups will be pre-tested before the procedure. 4. At the end of the massage, the test will be repeated.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peppermint oil (Experimental): Peppermint oil has an effect on menopausal symptoms
  Interventions: Other: peppermint oil
- Lemon oil (Experimental): Lemon oil has an effect on menopausal symptoms.
  Interventions: Other: Lemon oil
- almond oil (Placebo Comparator): Almond oil has an effect on menopausal symptoms.
  Interventions: Other: Almond oil

INTERVENTIONS:
Other: Lemon oil — Lemon oil with massage
  Arms: Lemon oil
Other: peppermint oil — peppermint oil with massage
  Arms: Peppermint oil
Other: Almond oil — Almond oil massage
  Arms: almond oil

SUMMARY:
Aromatherapy is "highly distilled herbs distilled to take advantage of their therapeutic properties".

is the science of using concentrated essential oils or essences".Essential oils or essences are obtained from various parts of plants (root, leaves, flowers, bark, fruit) and used therapeutically for physical and psychological well-being. The fact that aromatherapy is a noninvasive procedure and its ease of use allows for widespread use of aromatherapy. Aromatic oils can be applied in four basic ways. These include topical (tap, compress, or bath), internal (mouthwash, vaginal, or anal suppository), oral (with capsules or reconstitution in honey, alcohol, or diluent), and inhalation (direct or indirect, with or without steam, inhalation). ). Essential oils, which can be applied in various ways, can directly reach the neocortex part of the brain through connections extending from the limbic system to the hypothalamus via scent.

DETAILED DESCRIPTION:
As a result of the effect of aromatic oils on the central nervous system, relaxation, sedation or stimulating effects occur and the information flow reaching the brain with the stimulation of the central nervous system.

Thanks to this, the energy blockage in the body is broken and as a result, energy is released. With the balanced distribution of the energy flow to the relevant organs, the healing process is supported, and physical and mental well-being emerges . Aromatherapy is used in many health fields as well as women's health. Menopause is a process in which physiological, psychological and hormonal changes occur in the life of all women . The World Health Organization defines menopause as "the permanent cessation of menstruation with loss of ovarian activity" . In addition to physical symptoms such as hot flashes, sweating, headache, low libido, fatigue, sleep disorders, palpitations, which occur as a result of the decrease in estrogen and progesterone hormone secretion and its end over time, psychological symptoms such as anxiety, depression and mood disorders are frequently encountered . Due to the increase in the number of women in the menopausal period in the world, it is important to reduce menopausal complaints and improve women's health.Studies have shown that aromatherapy is a complementary method used in a wide variety of situations to reduce physiological and psychological symptoms . It is stated that menopausal symptoms decrease in women who smell lavender aroma during menopause . It is important that the symptoms seen during menopause, which is an important part of a woman's life, are reduced and that women can spend this process more comfortably. While the age at menopause is in the range of 50-51 years worldwide, it is reported that the age of menopause in our country is between the ages of 47-49 . From this point of view, women spend about one third of their lives during and after menopause. The trend towards traditional and complementary medicine is increasing day by day in our country. However, in addition to the widespread use of aromatherapy in the world, aromatherapy practices are not common in our country. Diluted and ready-to-use forms of aromatic oils are not only available in pharmacies and herbalists, but also a method that people are curious about and want to use. The fact that the cost of ready-to-use aromatic oils is cheaper than drugs and easily accessible will provide women with a treatment option in the light of new evidence in line with the conduct of the study. In studies in the literature, it is stated that lavender, rose, geranium, and citrus oils are massaged to women in the menopausal period and provide mental and physical relaxation. Therefore, in our study, the use of Peppermint and Lemon oils to reduce the symptoms of menopausal women and increase their psychosocial well-being. is planned. Peppermint (Mentha Piperita) oil has analgesic, immune system strengthening, antispasmodic, antipyretic, anti-nausea and vomiting, anesthetic, helps concentration, increases self-confidence and creative thoughts, and Lemon (Citrus Lemon) oil is analgesic, immune-enhancing, antipyretic. It is thought that it can help relieve the psychological and physiological complaints of women in the menopausal period due to its properties such as helping constipation, reducing nausea and vomiting, increasing sleep quality, relieving stress and antidepressant. For this reason, it is planned to use Peppermint and Lemon oils in our study.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing at least 1 of the menopausal symptoms (self-report),
* No respiratory disease such as asthma, bronchitis (self-report),
* Not allergic to the oils to be used (self-report),

Exclusion Criteria:

* Not experiencing menopausal complaints,
* Those who do not want to participate in the research

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — women in menopause
Enrollment: 90 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Menopause Symptoms Evaluation Scale | 1 year
  The original name of the scale is Menopause Rating Scale (MRS). The menopausal symptom rating scale (MSDS) was developed by Schneider et al. (2002) to measure the severity of menopausal symptoms. It was adapted into Turkish by Gürkan (2005). Menopause symptom assessment scale (MSDS) consists of 11 items. It is a Likert-type scale, and each item has options such as "None (0)", "Mild (1)", "Moderate (2)", "Severe (3)" and "Very Severe (4)". The total score of the scale is calculated by calculating the scores given for each item. A minimum of 0 points and a maximum of 44 points can be obtained from the scale. The increase in the total score obtained from the scale indicates the increase in the severity of the complaints. The Cronbach Alpha coefficient of the scale is 0.84.

CONTACTS AND LOCATIONS:
Overall Officials: HAFİZE DAĞ TÜZMEN, Principal Investigator — KTO Karatay University
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farahani MA, Afsargharehbagh R, Marandi F, Moradi M, Hashemi SM, Moghadam MP, Balouchi A. Effect of aromatherapy on cancer complications: A systematic review. Complement Ther Med. 2019 Dec;47:102169. doi: 10.1016/j.ctim.2019.08.003. Epub 2019 Aug 5. PMID 31779991
- [Background] Tanvisut R, Traisrisilp K, Tongsong T. Efficacy of aromatherapy for reducing pain during labor: a randomized controlled trial. Arch Gynecol Obstet. 2018 May;297(5):1145-1150. doi: 10.1007/s00404-018-4700-1. Epub 2018 Feb 3. PMID 29397442
- [Background] Santoro N, Epperson CN, Mathews SB. Menopausal Symptoms and Their Management. Endocrinol Metab Clin North Am. 2015 Sep;44(3):497-515. doi: 10.1016/j.ecl.2015.05.001. PMID 26316239
- [Background] Parry BL. Depressive history as a major predictor of postmenopausal depressive symptoms. Menopause. 2022 Jul 1;29(7):763-764. doi: 10.1097/GME.0000000000002027. No abstract available. PMID 35728014
- [Background] Lee J, Han Y, Cho HH, Kim MR. Sleep Disorders and Menopause. J Menopausal Med. 2019 Aug;25(2):83-87. doi: 10.6118/jmm.19192. Epub 2019 Aug 5. PMID 31497577
- [Background] Bansal R, Aggarwal N. Menopausal Hot Flashes: A Concise Review. J Midlife Health. 2019 Jan-Mar;10(1):6-13. doi: 10.4103/jmh.JMH_7_19. PMID 31001050
- [Background] Cramer H, Peng W, Lauche R. Yoga for menopausal symptoms-A systematic review and meta-analysis. Maturitas. 2018 Mar;109:13-25. doi: 10.1016/j.maturitas.2017.12.005. Epub 2017 Dec 6. PMID 29452777
- [Background] Johnson A, Roberts L, Elkins G. Complementary and Alternative Medicine for Menopause. J Evid Based Integr Med. 2019 Jan-Dec;24:2515690X19829380. doi: 10.1177/2515690X19829380. PMID 30868921
- [Background] Kazemzadeh R, Nikjou R, Rostamnegad M, Norouzi H. Effect of lavender aromatherapy on menopause hot flushing: A crossover randomized clinical trial. J Chin Med Assoc. 2016 Sep;79(9):489-92. doi: 10.1016/j.jcma.2016.01.020. Epub 2016 Jul 4. PMID 27388435
- [Background] Sanchez-Vidana DI, Ngai SP, He W, Chow JK, Lau BW, Tsang HW. The Effectiveness of Aromatherapy for Depressive Symptoms: A Systematic Review. Evid Based Complement Alternat Med. 2017;2017:5869315. doi: 10.1155/2017/5869315. Epub 2017 Jan 4. PMID 28133489
- [Background] Gurler M, Kizilirmak A, Baser M. The Effect of Aromatherapy on Sleep and Quality of Life in Menopausal Women with Sleeping Problems: A Non-Randomized, Placebo-Controlled Trial. Complement Med Res. 2020;27(6):421-430. doi: 10.1159/000507751. Epub 2020 Jun 9. PMID 32516765
- [Background] El Khoudary SR, Greendale G, Crawford SL, Avis NE, Brooks MM, Thurston RC, Karvonen-Gutierrez C, Waetjen LE, Matthews K. The menopause transition and women's health at midlife: a progress report from the Study of Women's Health Across the Nation (SWAN). Menopause. 2019 Oct;26(10):1213-1227. doi: 10.1097/GME.0000000000001424. PMID 31568098
- [Background] Taşkın L, editör. Doğum ve kadın sağlığı hemşireliği. Genişletilmiş XIII. Baskı. Ankara: Akadmisyen Tıp Kitabevi; 2019. p. 671-687
- [Background] Gözüyeşil E, Başer M. 2016.'' Menopozal dönemde yaşanan vazomotor yakınmaların günlük yaşam aktiviteleri üzerine etkisi'', Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi, 19(4):1-8.
- [Background] Türkiye İstatistik Kurumu. İstatistiklerle kadın, 2019. Türkiye İstatistik Kurumu Haber Bülteni. Sayı: 33732 Yayın Tarihi: 06.03.2020 1-5.
- [Background] Es-Haghee S, Shabani F, Hawkins J, Zareian MA, Nejatbakhsh F, Qaraaty M, Tabarrai M. The Effects of Aromatherapy on Premenstrual Syndrome Symptoms: A Systematic Review and Meta-Analysis of Randomized Clinical Trials. Evid Based Complement Alternat Med. 2020 Dec 21;2020:6667078. doi: 10.1155/2020/6667078. eCollection 2020. PMID 33414837
- [Background] Taavoni S, Darsareh F, Joolaee S, Haghani H. The effect of aromatherapy massage on the psychological symptoms of postmenopausal Iranian women. Complement Ther Med. 2013 Jun;21(3):158-63. doi: 10.1016/j.ctim.2013.03.007. Epub 2013 Apr 16. PMID 23642946
- [Background] Nikjou R, Kazemzadeh R, Asadzadeh F, Fathi R, Mostafazadeh F. The Effect of Lavender Aromatherapy on the Symptoms of Menopause. J Natl Med Assoc. 2018 Jun;110(3):265-269. doi: 10.1016/j.jnma.2017.06.010. Epub 2017 Aug 18. PMID 29778129
- [Background] Hur MH, Yang YS, Lee MS. Aromatherapy massage affects menopausal symptoms in korean climacteric women: a pilot-controlled clinical trial. Evid Based Complement Alternat Med. 2008 Sep;5(3):325-8. doi: 10.1093/ecam/nem027. PMID 18830459
- [Background] Abbaspoor Z, Siahposh A, Javadifar N, Faal Siahkal S, Mohaghegh Z, Sharifipour F. The Effect of Citrus Aurantium Aroma on the Sleep Quality in Postmenopausal Women: A Randomized Controlled Trial. Int J Community Based Nurs Midwifery. 2022 Apr;10(2):86-95. doi: 10.30476/IJCBNM.2021.90322.1693. PMID 35372632
- [Background] Darsareh F, Taavoni S, Joolaee S, Haghani H. Effect of aromatherapy massage on menopausal symptoms: a randomized placebo-controlled clinical trial. Menopause. 2012 Sep;19(9):995-9. doi: 10.1097/gme.0b013e318248ea16. PMID 22549173
- [Background] Tsai J, Chung YC, Chen FP, Yeh ML. [Effect of Aromatherapy on Menopausal Symptoms, Heart Rate Variability, and Sleep Quality in Women]. Hu Li Za Zhi. 2020 Feb;67(1):44-54. doi: 10.6224/JN.202002_67(1).07. Chinese. PMID 31960396
- [Background] Dos Reis Lucena L, Dos Santos-Junior JG, Tufik S, Hachul H. Lavender essential oil on postmenopausal women with insomnia: Double-blind randomized trial. Complement Ther Med. 2021 Jun;59:102726. doi: 10.1016/j.ctim.2021.102726. Epub 2021 Apr 24. PMID 33905827
- [Derived] Doner SI, Dag Tuzmen H, Duran B, Sunar F. The effect of aromatherapy massage with lemon and peppermint essential oil on menopausal symptoms: A double-blinded, randomized placebo controlled clinical trial. Explore (NY). 2024 May-Jun;20(3):313-318. doi: 10.1016/j.explore.2023.09.001. Epub 2023 Sep 13. PMID 37743153
- See also: World Health Organization (1981). Research on the menapouse. Available date: 16.08.2022 — http://apps.who.int/iris/bitstream/handle/10665/41526/WHO_TRS_670.pdf;jsessionid=90771D3E84AEA4AEC1439F900E135632?sequence=1